CLINICAL TRIAL: NCT05408039
Title: A Prospective, Non-interventional, Longitudinal Study of the Treatment Journey of Adult Patients With Hyperkalemia
Brief Title: Tracking Treatment Pathways in Adult Patients With Hyperkalemia.
Acronym: TRACK
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9480R00048
Record Dates: First submitted 2022-05-18; First posted 2022-06-07 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hyperkalemia
Keywords: Treatment pathways,; Hyperkalemia,; High level of Serum potassium.; Treatment rationale,; Treatment objective,; Treatment expectations,; Heart failure and; Chronic kidney disease.
MeSH Terms: conditions — Hyperkalemia; Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Not applicable. No Samples Retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to increase the understanding of Hyperkalemia (HK) management, treatment patterns, and the treatment decision-making process for the management of patients with HK over a period of up to 12 months. The generation of real-world evidence (RWE) to understand the treatment management decision rationale and to prospectively describe patient characteristics, treatment management patterns among patients with HK is of importance to improve adherence to guidelines and improve patient care.

The primary objective:

• Describe HK management decisions, their rationale and treatment expectations.

The secondary objective:

• Describe baseline characteristics and longitudinal clinical variables in patients with HK.

The exploratory objective:

• Describe patient awareness and satisfaction with their HK treatment management across the study period.

DETAILED DESCRIPTION:
This study is a multinational, observational, prospective, longitudinal, cohort study that will include primary and secondary data collection. Secondary data, collected as per routine clinical practice will be extracted from electronic health records (EHR) and manually entered into the electronic case report form (eCRF). Primary data will be collected directly from patients and Health Care Providers (HCPs). Prospective data collection will be performed for a period of 12 months and will include data collection at baseline, that is, the date of enrollment, and at 3-, 6-, 9-, and 12-months following baseline. The data collection timepoints in this study is irrespective of when the patient's medical visits are scheduled. There are no study specific patient visits mandated by protocol and study may be fully virtual.

ELIGIBILITY:
Patients meeting all the following inclusion criteria will be eligible for inclusion into the study:

1. Age ≥18 years on the date of signing informed consent
2. HK with serum potassium (K+) level(s) greater than 5.0 mmol/L, collected during Standard of Care, within 21 days prior to the date of enrollment*
3. Provision of signed and dated informed consent

(*enrollment in study is defined as the date of Informed consent and confirmation of study eligibility, whichever occurs later).

Patients will be excluded from the study if they meet any of the following criteria:

1. Concurrent participation in any trial that includes the use of K+ binders as an investigational medicinal product (IMP)
2. Patients with pseudohyperkalemia
3. A life expectancy of less than six months, based on physician judgement
4. Acute causes of HK such as infections and/or trauma to be determined by the principal investigator
5. Scheduled renal transplant
6. Involvement in the planning and/or conduct of the study

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with established HK (K+ levels >5.0 mmol/L) at selected sites distributed across USA and Europe will be recruited by the principal investigators to participate in the study.
  This is a non-interventional study. As such, patients will undergo clinical assessments and receive standard medical care as determined by their treating physicians. Patients will not receive any experimental disease management intervention or experimental treatment because of their participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1331 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Description of change in HK management decision at 3 month intervals. | Up to 12 months following enrolment.
Description of HK management objective(s) decision at 3 month intervals. | Up to 12 months following enrolment.
Description of expected HK management duration decision at 3 month intervals. | Up to 12 months following enrolment.

SECONDARY OUTCOMES:
Change in time to K+ normalization at 3 month intervals. | Up to 12 months following enrolment.
Description of HK recurrence frequency. | Up to 12 months following enrolment.
Description of average dose of Renin angiotensin aldosterone system inhibitor (RAASi) therapy. | Up to 12 months following enrolment.
Change in time to achieve target dose of Renin angiotensin aldosterone system inhibitor (RAASi) therapy at 3 month intervals. | Up to 12 months following enrolment.
Description of occurrences of HK complications such as arrythmia, muscle weakness, and metabolic acidosis. | Up to 12 months following enrolment.
Description of Healthcare resource utilization (HCRU). | Up to 12 months following enrolment.

OTHER OUTCOMES:
Description of change in awareness and satisfaction to HK management by patient reported outcome (PRO) at 3 month intervals. | Up to 12 months following enrolment.
  Functional Assessment of Chronic Illness Therapy Treatment Satisfaction-General (FACIT-TS-G) and bespoke questions on dietary recommendations.

CONTACTS AND LOCATIONS:
Locations (74):
- United States (17):
  - Research Site, Huntsville, Alabama
  - Research Site, La Jolla, California
  - Research Site, Rancho Cucamonga, California
  - Research Site, New Haven, Connecticut
  - Research Site, Nampa, Idaho
  - Research Site, Hinsdale, Illinois
  - Research Site, Princeton, New Jersey
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Abington, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Edinburg, Texas
  - Research Site, Houston, Texas
  - Research Site, Burlington, Vermont
- Germany (9):
  - Research Site, Bad Krozingen
  - Research Site, Berlin
  - Research Site, Coburg
  - Research Site, Dresden
  - Research Site, Fulda
  - Research Site, Göttingen
  - Research Site, Halle
  - Research Site, Papenburg
  - Research Site, Stuttgart
- Italy (17):
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Parma
  - Research Site, Pisa
  - Research Site, Rome
  - Research Site, Rozzano
  - Research Site, San Giovanni Rotondo
  - Research Site, Sassari
  - Research Site, Trieste
- Spain (15):
  - Research Site, Badalona
  - Research Site, Barcelona
  - Research Site, El Ejido
  - Research Site, El Palmar
  - Research Site, Ferrol
  - Research Site, Gij N
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Ja N
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Salamanca
  - Research Site, San Sebasti N de Los Reyes
  - Research Site, Sant Joan Despí
  - Research Site, Zaragoza
- United Kingdom (16):
  - Research Site, Ashford
  - Research Site, Barnet
  - Research Site, Barnstaple
  - Research Site, Birkenhead
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Calow
  - Research Site, Dorchester
  - Research Site, Headington
  - Research Site, High Heaton/Newcastle Upon Tyn
  - Research Site, Hull
  - Research Site, Kogarah
  - Research Site, London
  - Research Site, Preston
  - Research Site, Salford
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Hsia J, Shivappa N, Bakhai A, Bover J, Butler J, Ferraro PM, Fried L, Schneider MP, Tangri N, Winkelmayer WC, Bishop M, Chen H, Sundin AK, Bonaca MP. Design and cohort characteristics of TRACK, a prospective study of hyperkalaemia management decision-making. Clin Kidney J. 2024 Sep 30;17(10):sfae295. doi: 10.1093/ckj/sfae295. eCollection 2024 Oct. PMID 39464260
- See also: D9480R00048 CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9480R00048&attachmentIdentifier=c207a9a1-995e-4c2d-a480-9e70368a33ca&fileName=D9480R00048_CSR_Synopsis_Redacted.pdf&versionIdentifier=